CLINICAL TRIAL: NCT00904163
Title: Characteristics of Adult Patients With Recessive Dystrophic Epidermolysis Bullosa
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alfred Lane, Professor of Dermatology and Pediatrics, Stanford University
Other Study IDs: SU-04232009-2383
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies, serum

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) is a severe inherited blistering disease caused by the absence of type VII collagen. Patients with RDEB develop large, severely painful blisters and open wounds from minor trauma to their skin. We are screening RDEB subjects to determine additional characteristics of patients who survive to adulthood.

ELIGIBILITY:
Inclusion Criteria:1. Clinical diagnosis of RDEB by local dermatologist. 2. 18 years of age or more and willing to give consent. Exclusion Criteria:1. Medical instability limiting ability to travel to Stanford University Medical Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years of age or older) with RDEB diagnosis by a local dermatologist, who can travel to Stanford University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred T Lane, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States